CLINICAL TRIAL: NCT05097781
Title: Evaluating the Efficacy of Local Radiotherapy in Combination With Immunotherapy in Advanced Solid Tumors: a Phase II Prospective Clinical Study
Brief Title: Local Radiotherapy in Combination With Immunotherapy in Advanced Solid Tumors Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jiayi Chen, Chief of Department of Radiation Oncology, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RuijinHDR
Record Dates: First submitted 2021-07-28; First posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Local irradiation + immunotherapy
  Interventions: Drug: PD-1 blocking antibody

INTERVENTIONS:
Drug: PD-1 blocking antibody — All patients with more than one distant metastatic lesions will accept at least one site of radiotherapy and PD-1 blockade at the same time.
  Other Names: irradiation

SUMMARY:
This is a phase II study to observe efficacy of combining local radiotherapy with PD-1blockade in patients with advanced solid tumors. All patients will accept at least one site of radiotherapy together with PD-1 blockade. The study will evaluate changes of unirradiated and irradiated lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients 18-75 years old with the right to make medical decisions
2. Signed informed consent form
3. ECOG score of 0-2
4. Clear pathological diagnosis of the primary site
5. Multiple distant metastases
6. Stable assessment of brain metastases after treatment can be enrolled (more than 6 weeks)
7. Bone metastases combined with soft tissue mass formation can be enrolled
8. imaging with ≥ 2 clearly assessable lesions (bone metastases alone without soft tissue mass formation, brain metastases not as target lesions)
9. expected survival ≥ 6 months
10. Progression after ≥ 1 prior line of therapy regimen with no standard treatment regimen or intolerable toxicities, including all three of the following:

    1. Patients must have failed to respond to at least one prior standard of care regimen
    2. The patient must not have a conventional treatment option that is clinically proven to provide long-term control of the disease and the patient refuses other conventional treatment options
    3. The patient is intolerant to the toxic side effects of the standard treatment regimen
11. No prior immunotherapy history
12. Time to last systemic therapy (including monoclonal antibodies) ≥ 4 weeks
13. Previous radiotherapy to non-target sites with other evaluable lesions can be enrolled
14. Laboratory examination indexes meet the following requirements: WBC ≥ 3×109/L, ANC ≥ 2.0×109/L, PLT ≥ 80×109/L, Hb ≥ 80g/L (according to the normal standards of the central laboratory department); liver function: total bilirubin, ALT and AST are ≤ 1.5xUNL (upper limit of normal value); AST (SGOT)/ALT (SGPT) ≤ 2.5xUNL (upper limit of normal value) ALT (SGPT) ≤ 2.5 x IULN (upper limit of normal value); renal function: Cr≦1.5xUNL (upper limit of normal value), and creatinine clearance rate≧60ml/min; thyroid function T3, T4 within normal range (hypothyroidism can be supplemented with oral thyroxine); cardiac function: cardiac protein three and pro-BNP within normal range, no previous Adrenal function: normal cortisol secretion function or correctable by endocrine assessment
15. HBV infected patients with HBV-DNA copy number less than 500 IU/ml
16. No history of other malignancies within 5 years (except skin basal cell carcinoma)

Exclusion Criteria:

1. Uncontrolled brain metastases (stabilization time <6 weeks)
2. Bone metastases alone without clear soft tissue mass formation
3. Bone marrow infiltration
4. Presence of clinical factors (e.g., bleeding, active infection, or psychiatric factors) that the investigator determines may interfere with the completion of the study process
5. Inability to administer radiotherapy due to organ-threatening or other factors as assessed by the investigator
6. Patients requiring long-term maintenance steroid therapy (including oral, intravenous use); topical use or inhalation may be included in the study
7. Prior autoimmune disease or active disease [e.g., including but not limited to inflammatory bowel disease [IBD], rheumatoid arthritis, autoimmune hepatitis, systemic sclerosis (scleroderma and its variants), systemic lupus erythematosus, autoimmune vasculitis, autoimmune neuropathy (e.g., Guillain-Barre syndrome)], vitiligo and correctable endocrine deficiencies such as thyroid hypofunction, physiological cortisol hypersecretion may be included in the study and are not considered as exclusion criteria.
8. history of active tuberculosis or non-infectious pneumonia or any clinical evidence
9. Active viral hepatitis with HBV DNA > 500 IU/ml
10. Immunodeficiency syndrome
11. comorbid serious medical disorders with concomitant diseases or conditions affecting the normal enrollment of the patient or safety during the study
12. previous immunotherapy for other tumors
13. History of other malignancies within 5 years (except cured basal cell carcinoma of the skin);
14. Pregnant or lactating women;
15. Unable or unwilling to sign the informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-03-21 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed at least 4 weeks
  The proportion of patients with a tumor volume reduction of 30% lasting for at least 4 weeks，and is the sum of the proportion of complete remission (CR) and partial remission (PR)
non-irradiated lesion control rate(NRCR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  The percentage of non-irradiated target lesions with CR/PR or SD

SECONDARY OUTCOMES:
Progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  The time from enrollment to disease progression or death from any cause
Overall survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  The time from enrollment to death from any cause
Rate of side effects | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  ≥ grade 3 adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Jiayi Chen, MD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No